CLINICAL TRIAL: NCT01167335
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Exploratory Study to Assess the Antiepileptic Activity of BGG492 Given Orally as Adjunctive Treatment in Patients With Refractory Partial Onset Seizures
Brief Title: Evaluate the Efficacy of BGG492 as Adjunctive Treatment in Patients With Refractory Partial Onset Seizures
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGG492A2211; 2010-018766-23 (EudraCT Number)
Record Dates: First submitted 2010-06-25; First posted 2010-07-22 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Partial Onset Seizures
Keywords: partial onset seizure; seizure frequency; nervous system diseases; central nervous system diseases; CNS; brain diseases; neurologic manifestations; adjunctive treatment; AEDs; antiepileptic drug
MeSH Terms: conditions — Nervous System Diseases; Central Nervous System Diseases; Brain Diseases; Neurologic Manifestations | interventions — selurampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BGG492 (Experimental)
  Interventions: Drug: BGG492
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGG492
  Arms: BGG492
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of BGG492 as adjunctive treatment in patients with refractory partial onset seizures

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 50 kg (110 lb) of weight
* A diagnosis of epilepsy (≥ 2 years prior to screening) with partial seizures with or without secondarily generalized seizures
* Uncontrolled partial seizures despite having been treated with at least two different AEDs within the last 2 years prior to screening.
* Treated with a stable dose of 1-2 AEDs
* At least 4 partial seizures during the 4-week baseline period and at least 4 partial seizures during the 4 weeks prior to the baseline period.
* No 28-day seizure-free period during the 8 weeks preceding randomization
* Positive biomarker screening

Exclusion Criteria:

* Presence of only non-motor simple partial seizures
* History of psychogenic seizures
* Absences, myoclonic seizures e.g. in the context of primary generalized epilepsy;
* Previous history of Lennox-Gastaut syndrome
* Pregnant or nursing (lactating) women
* Status epilepticus or seizure clusters, according to the judgement of the investigator, occurring within 52 weeks prior to randomization

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Seizure counts, documenting the percent change in seizure frequency of BGG492 in the maintenance period. | 28 days

SECONDARY OUTCOMES:
Responder rate: analysis of patients with a 50% or greater reduction in seizure frequency of BGG492 during the maintenance period. | 28 days
Safety and tolerability of BGG492 compared to placebo evaluated by continuous adverse event monitoring and assessment of vital signs and ECGs at each visit and laboratory assessments every 2 to 4 weeks | 12 weeks
Pharmacokinetic profile of BGG492 including plasma concentrations of BGG492 at each dose level and derived variables including AUC (area under the curve), Cmax (maximum plasma concentration), Tmax (time to maximum concentration), T1/2 (half life.) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (3):
  - University of South Alabama, Mobile, Alabama
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Epilepsy Care Specialists, S.C., Milwaukee, Wisconsin
- Austria (3):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
  - Novartis Investigational Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Duffel
  - Novartis Investigative Site, Ottignies
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- India (4):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Dehli, New Delhi
  - Novartis Investigative Site, Jaipur
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Kaunas, Lithuania
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Barcelona, Spain